CLINICAL TRIAL: NCT02044796
Title: A Phase 1/2 Trial of G-CSF, Cladribine, Cytarabine, and Dose-Escalated Mitoxantrone (G-CLAM) in Adults With Newly Diagnosed or Relapsed/Refractory Acute Myeloid Leukemia (AML) or High-Risk Myelodysplastic Syndromes (MDS)
Brief Title: Filgrastim, Cladribine, Cytarabine, and Mitoxantrone Hydrochloride in Treating Patients With Newly Diagnosed or Relapsed/Refractory Acute Myeloid Leukemia or High-Risk Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2734.00; NCI-2013-02465 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2734.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2020-01-10 (Actual); Status verified 2019-12

CONDITIONS: Acute Biphenotypic Leukemia; de Novo Myelodysplastic Syndrome; Previously Treated Myelodysplastic Syndrome; Recurrent Adult Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute; Leukemia, Myeloid, Acute | interventions — Cladribine; Cytarabine; Filgrastim; Granulocyte Colony-Stimulating Factor; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (filgrastim, mitoxantrone, cladribine, cytarabine) (Experimental): INDUCTION CHEMOTHERAPY (G-CLAM): Patients receive G-CLAM chemotherapy comprising filgrastim SC daily on days 0-5, mitoxantrone hydrochloride IV over 60 minutes on days 1-3, cladribine IV over 2 hours daily on days 1-5, and cytarabine IV over 2 hours daily on days 1-5. Patients achieving CRi, partial remission, or persistent disease may receive a second course of induction chemotherapy. Patients achieving CR or CRp may continue on to Consolidation Chemotherapy.
  CONSOLIDATION CHEMOTHERAPY (G-CLA): Beginning within 6 weeks of achieving CR/CRp/CRi, patients receive G-CLA comprising filgrastim SC on days 0-5, cladribine IV over 2 hours daily on days 1-5, and cytarabine IV over 2 hours daily on days 1-5. Treatment continues for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cladribine; Drug: Cytarabine; Biological: Filgrastim; Other: Laboratory Biomarker Analysis; Drug: Mitoxantrone Hydrochloride

INTERVENTIONS:
Drug: Cladribine — Given IV
  Other Names: 2-CdA; 2CDA; CdA; Cladribina; Leustat; Leustatin; Leustatine; RWJ-26251
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Biological: Filgrastim — Given SC
  Other Names: Filgrastim XM02; Filgrastim-sndz; G-CSF; Neupogen; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tbo-filgrastim; Tevagrastim; Zarxio
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Mitoxantrone Hydrochloride — Given IV
  Other Names: CL 232315; DHAD; DHAQ; Dihydroxyanthracenedione Dihydrochloride; Mitoxantrone Dihydrochloride; Mitoxantroni Hydrochloridum; Mitozantrone Hydrochloride; Mitroxone; Neotalem; Novantrone; Onkotrone; Pralifan

SUMMARY:
This phase I/II trial studies the side effects and best dose of mitoxantrone hydrochloride when given together with filgrastim, cladribine, and cytarabine and to see how well they work in treating patients with acute myeloid leukemia or high-risk myelodysplastic syndromes that is newly diagnosed, has returned, or does not respond to treatment. Drugs used in chemotherapy, such as filgrastim, cladribine, cytarabine, and mitoxantrone hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Estimate the maximum tolerated dose (MTD) of dose-intensified mitoxantrone hydrochloride (mitoxantrone) as part of the filgrastim (G-CSF), cladribine, cytarabine, mitoxantrone hydrochloride (G-CLAM) regimen separately for adults with newly diagnosed acute myeloid leukemia (AML) and those with relapsed/refractory AML receiving first or greater salvage therapy.

SECONDARY OBJECTIVES:

I. To determine, within the limits of a phase 1/2 study, disease response and duration of remission separately for patients with newly diagnosed and relapsed/refractory AML.

II. To describe, within the limits of a phase 1/2 study, the toxicity profile of the study regimen separately for patients with newly diagnosed and relapsed/refractory AML.

OUTLINE: This is a phase I, dose-escalation study of mitoxantrone hydrochloride followed by phase II study.

INDUCTION CHEMOTHERAPY (G-CLAM): Patients receive G-CLAM chemotherapy comprising filgrastim subcutaneously (SC) daily on days 0-5, mitoxantrone hydrochloride intravenously (IV) over 60 minutes on days 1-3, cladribine IV over 2 hours daily on days 1-5, and cytarabine IV over 2 hours daily on days 1-5. Patients achieving complete remission with incomplete peripheral blood count recovery (CRi), partial remission, or persistent disease may receive a second course of induction chemotherapy. Patients achieving complete remission (CR) or CR with incomplete platelet count recovery (CRp) may continue on to Consolidation Chemotherapy.

CONSOLIDATION CHEMOTHERAPY (G-CLA): Beginning within 6 weeks of achieving CR/CRp/CRi, patients receive G-CLA comprising filgrastim SC on days 0-5, cladribine IV over 2 hours daily on days 1-5, and cytarabine IV over 2 hours daily on days 1-5. Treatment continues for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* For patients with newly diagnosed disease: diagnosis of "high-risk" myelodysplastic syndrome (MDS) (>= 10% blasts) or AML other than acute promyelocytic leukemia (APL) with t(15;17)(q22;q12) or variants according to the 2008 World Health Organization (WHO) classification; for patients with relapsed/refractory disease: prior diagnosis of "high-risk" MDS or non-APL AML, with relapsed/refractory disease according to standard criteria requiring first or subsequent salvage therapy; patients with biphenotypic AML are eligible
* Outside diagnostic material is acceptable as long as peripheral blood and/or bone marrow slides are reviewed at the study institution; flow cytometric analysis of peripheral blood and/or bone marrow should be performed according to institutional practice guidelines
* For patients with relapsed/refractory disease: patients with prior autologous or allogeneic hematopoietic cell transplantation (HCT) for MDS/AML are eligible if relapse occurs provided symptoms of graft-versus host disease are well controlled with stable use of immunosuppressive agents
* Treatment-related mortality (TRM) score =< 6.9 as calculated with simplified model
* The use of hydroxyurea prior to study registration is allowed; patients with symptoms/signs of hyperleukocytosis or white blood cell (WBC) > 100,000/uL can be treated with leukapheresis or may receive up to 2 doses of cytarabine (up to 500 mg/m^2/dose) prior to enrollment
* For patients with relapsed/refractory disease: patients may have previously received chemotherapy with a mitoxantrone- or cladribine-based regimen for MDS or AML; if that patient has received G-CLAM before and has been sensitive to this regimen, eligibility will be determined on a case-by-case basis by the study principal investigator (PI)
* Should be off any active systemic therapy for AML with the exception of hydroxyurea for at least 14 days prior to study registration unless patient has rapidly progressive disease, and all grade 2-4 non-hematologic toxicities should have resolved
* Bilirubin =< 2.5 x institutional upper limit of normal (IULN) unless elevation is thought to be due to hepatic infiltration by AML, Gilbert's syndrome, or hemolysis (assessed within 14 days prior to study day 0)
* Serum creatinine =< 2.0 mg/dL (assessed within 14 days prior to study day 0)
* Left ventricular ejection fraction >= 45%, assessed within 3 months prior to study day 0, e.g. by multi gated acquisition scan (MUGA) scan or echocardiography, or other appropriate diagnostic modality and no clinical evidence of congestive heart failure; if the patient had anthracycline-based therapy since the most recent cardiac assessment, cardiac evaluation should be repeated if there is clinical or radiographic suspicion of cardiac dysfunction, or if the previous cardiac assessment was abnormal
* Women of childbearing potential and men must agree to use adequate contraception
* Provide written informed consent

Exclusion Criteria:

* Myeloid blast crisis of chronic myeloid leukemia (CML), unless patient is not considered candidate for tyrosine kinase inhibitor treatment
* Concomitant illness associated with a likely survival of < 1 year
* Active systemic fungal, bacterial, viral, or other infection, unless disease is under treatment with anti-microbials and/or controlled or stable (e.g. if specific, effective therapy is not available/feasible or desired [e.g. chronic viral hepatitis, human immunodeficiency virus (HIV)]); patient needs to be clinically stable as defined as being afebrile and hemodynamically stable for 24 hours; patients with fever thought to be likely secondary to leukemia are eligible
* Known hypersensitivity to any study drug
* Pregnancy or lactation
* Treatment with any other investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2014-01-23 (Actual); Primary Completion 2018-03-09 (Actual); Study Completion 2018-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roland Walter, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Newly Diagnosed Group Mitoxantrone Hydrochloride 12 mg/m^2; Newly Diagnosed Group Mitoxantrone Hydrochloride 14 mg/m^2; Newly Diagnosed Group Mitoxantrone Hydrochloride 16 mg/m^2; Newly Diagnosed Group Mitoxantrone Hydrochloride 18mg/m^2; Relapsed/Refractory Group Mitoxantrone Hydrochloride 12 mg/m^2; Relapsed/Refractory Group Mitoxantrone Hydrochloride 14 mg/m^2; Relapsed/Refractory Group Mitoxantrone Hydrochloride 16 mg/m^2; Relapsed/Refractory Group Mitoxantrone Hydrochloride 18 mg/m^2; Phase 2 Newly Diagnosed Group 18 mg/m^2; Phase 2 Relapsed/Refractory Group 16 mg/m^2: INDUCTION CHEMOTHERAPY (G-CLAM): Patients receive G-CLAM chemotherapy comprising filgrastim SC daily on days 0-5, mitoxantrone hydrochloride IV over 60 minutes on days 1-3, cladribine IV over 2 hours daily on days 1-5, and cytarabine IV over 2 hours daily on days 1-5. Patients achieving CRi, partial remission, or persistent disease may receive a second course of induction chemotherapy. Patients achieving CR or CRp may continue on to Consolidation Chemotherapy.
  CONSOLIDATION CHEMOTHERAPY (G-CLA): Beginning within 6 weeks of achieving CR/CRp/CRi, patients receive G-CLA comprising filgrastim SC on days 0-5, cladribine IV over 2 hours daily on days 1-5, and cytarabine IV over 2 hours daily on days 1-5. Treatment continues for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Cladribine: Given IV
  Cytarabine: Given IV
  Filgrastim: Given SC
  Laboratory Biomarker Analysis: Correlative studies
  Mitoxantrone Hydrochloride: Given IV
Period: Overall Study
Arm/Group | Newly Diagnosed Group Mitoxantrone Hydrochloride 12 mg/m^2 | Newly Diagnosed Group Mitoxantrone Hydrochloride 14 mg/m^2 | Newly Diagnosed Group Mitoxantrone Hydrochloride 16 mg/m^2 | Newly Diagnosed Group Mitoxantrone Hydrochloride 18mg/m^2 | Relapsed/Refractory Group Mitoxantrone Hydrochloride 12 mg/m^2 | Relapsed/Refractory Group Mitoxantrone Hydrochloride 14 mg/m^2 | Relapsed/Refractory Group Mitoxantrone Hydrochloride 16 mg/m^2 | Relapsed/Refractory Group Mitoxantrone Hydrochloride 18 mg/m^2 | Phase 2 Newly Diagnosed Group 18 mg/m^2 | Phase 2 Relapsed/Refractory Group 16 mg/m^2
Started | 9 | 9 | 9 | 6 | 10 | 6 | 6 | 4 | 106 | 34
Completed | 9 | 9 | 9 | 6 | 10 | 6 | 6 | 4 | 106 | 34
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Newly Diagnosed; Relapsed/Refractory Group: INDUCTION CHEMOTHERAPY (G-CLAM): Patients receive G-CLAM chemotherapy comprising filgrastim SC daily on days 0-5, mitoxantrone hydrochloride IV over 60 minutes on days 1-3, cladribine IV over 2 hours daily on days 1-5, and cytarabine IV over 2 hours daily on days 1-5. Patients achieving CRi, partial remission, or persistent disease may receive a second course of induction chemotherapy. Patients achieving CR or CRp may continue on to Consolidation Chemotherapy.
  CONSOLIDATION CHEMOTHERAPY (G-CLA): Beginning within 6 weeks of achieving CR/CRp/CRi, patients receive G-CLA comprising filgrastim SC on days 0-5, cladribine IV over 2 hours daily on days 1-5, and cytarabine IV over 2 hours daily on days 1-5. Treatment continues for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Cladribine: Given IV
  Cytarabine: Given IV
- Total: Total of all reporting groups
Arm/Group | Newly Diagnosed | Relapsed/Refractory Group | Total
Number analyzed (Participants) | 139 | 60 | 199
Age, Continuous [Mean (Full Range); unit: years] | 58.1 [18 to 80] | 58.2 [33 to 76] | 58.1 [18 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 25 | 84
  Male | 80 | 35 | 115
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 7 | 3 | 10
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  Black or African American | 6 | 1 | 7
  White | 112 | 52 | 164
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities of Mitoxantrone (Phase I, Dose Level 4)
Description: Defined as the highest dose studied in which the incidence of dose-limiting toxicity is < 33%, graded according to NCI Common Terminology Criteria for Adverse Events version 4.0
Time Frame: Up to day 45 after start of induction chemotherapy
Measure: Count of Participants; unit: Participants
Groups:
- Newly Diagnosed Group; Relapsed/Refractory Group: INDUCTION CHEMOTHERAPY (G-CLAM): Patients receive G-CLAM chemotherapy comprising filgrastim SC daily on days 0-5, mitoxantrone hydrochloride IV over 60 minutes on days 1-3, cladribine IV over 2 hours daily on days 1-5, and cytarabine IV over 2 hours daily on days 1-5. Patients achieving CRi, partial remission, or persistent disease may receive a second course of induction chemotherapy. Patients achieving CR or CRp may continue on to Consolidation Chemotherapy.
  CONSOLIDATION CHEMOTHERAPY (G-CLA): Beginning within 6 weeks of achieving CR/CRp/CRi, patients receive G-CLA comprising filgrastim SC on days 0-5, cladribine IV over 2 hours daily on days 1-5, and cytarabine IV over 2 hours daily on days 1-5. Treatment continues for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Cladribine: Given IV
  Cytarabine: Given IV
  Filgrastim: Given SC
  Laboratory Biomarker Analysis: Correlative studies
  Mitoxantrone Hydrochloride: Given IV
Arm/Group | Newly Diagnosed Group | Relapsed/Refractory Group
Number analyzed (Participants) | 6 | 4
Participants | 1 | 2

2. Primary Outcome: Minimal Residual Disease Negative Complete Remission Rate in Patients With Newly Diagnosed Disease (Phase II)
Description: Remission Rate defined as Recist Category of Complete Resposne (CR) Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size(<10 mm short axis).
Time Frame: Up to day 45 after start of second course of induction chemotherapy
Measure: Count of Participants; unit: Participants
Groups:
- Relapsed/Refractory: INDUCTION CHEMOTHERAPY (G-CLAM): Patients receive G-CLAM chemotherapy comprising filgrastim SC daily on days 0-5, mitoxantrone hydrochloride IV over 60 minutes on days 1-3, cladribine IV over 2 hours daily on days 1-5, and cytarabine IV over 2 hours daily on days 1-5. Patients achieving CRi, partial remission, or persistent disease may receive a second course of induction chemotherapy. Patients achieving CR or CRp may continue on to Consolidation Chemotherapy.
  CONSOLIDATION CHEMOTHERAPY (G-CLA): Beginning within 6 weeks of achieving CR/CRp/CRi, patients receive G-CLA comprising filgrastim SC on days 0-5, cladribine IV over 2 hours daily on days 1-5, and cytarabine IV over 2 hours daily on days 1-5. Treatment continues for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Cladribine: Given IV
  Cytarabine: Given IV
  Filgrastim: Given SC
  Laboratory Biomarker Analysis: Correlative studies
  Mitoxantrone Hydrochloride: Given IV
Arm/Group | Newly Diagnosed Group | Relapsed/Refractory
Number analyzed (Participants) | 112 | 40
Participants | 95 | 22

3. Secondary Outcome: Overall Survival (Phase II)
Description: Number of subjects that have survived
Time Frame: From date of randomization until the date of death from any cause, assessed up to 12 months
Measure: Number; unit: Participants
Arm/Group | Phase 2 Newly Diagnosed Group 18 mg/m^2 | Phase 2 Relapsed/Refractory Group 16 mg/m^2
Number analyzed (Participants) | 106 | 34
Participants | 66 | 13

4. Secondary Outcome: Remission Rate (Complete Remission and Complete Remission With Incomplete Platelet Count Recovery) of This Regimen in Patients With Relapsed/Refractory Disease (Phase II)
Time Frame: Up to 5 years
Population: Per the protocol, the 6 patients enrolled in the Phase 1 portion and treated at the MTD dose (16 mg/m^2) were included in the analysis of the Phase 2 remission rate.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Relapsed/Refractory Group 16 mg/m^2
Number analyzed (Participants) | 40
Participants | 24

ADVERSE EVENTS:
Time Frame: All-Cause Mortality assessed for up to 12 months; Serious and Other Adverse Events assessed for up to 1 month after treatment concluded
Groups:
- Newly Diagnosed Group Mitoxantrone Hydrochloride 18 mg/m^2; Relapsed/Refractory Group Mitoxantrone Hydrochloride 12 mg/m^2; Relapsed/Refractory Group Mitoxantrone Hydrochloride 14 mg/m^2; Relapsed/Refractory Group Mitoxantrone Hydrochloride 16 mg/m^2; Relapsed/Refractory Group Mitoxantrone Hydrochloride 18 mg/m^2; Phase 2 Newly Diagnosed Group 18 mg/m^2; Phase 2 Relapsed/Refractory Group 16 mg/m^2: INDUCTION CHEMOTHERAPY (G-CLAM): Patients receive G-CLAM chemotherapy comprising filgrastim SC daily on days 0-5, mitoxantrone hydrochloride IV over 60 minutes on days 1-3, cladribine IV over 2 hours daily on days 1-5, and cytarabine IV over 2 hours daily on days 1-5. Patients achieving CRi, partial remission, or persistent disease may receive a second course of induction chemotherapy. Patients achieving CR or CRp may continue on to Consolidation Chemotherapy.
  CONSOLIDATION CHEMOTHERAPY (G-CLA): Beginning within 6 weeks of achieving CR/CRp/CRi, patients receive G-CLA comprising filgrastim SC on days 0-5, cladribine IV over 2 hours daily on days 1-5, and cytarabine IV over 2 hours daily on days 1-5. Treatment continues for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Cladribine: Given IV
  Cytarabine: Given IV
  Filgrastim: Given SC
  Laboratory Biomarker Analysis: Correlative studies
  Mitoxantrone Hydrochloride: Given IV
Arm/Group | Newly Diagnosed Group Mitoxantrone Hydrochloride 12 mg/m^2 | Newly Diagnosed Group Mitoxantrone Hydrochloride 14 mg/m^2 | Newly Diagnosed Group Mitoxantrone Hydrochloride 16 mg/m^2 | Newly Diagnosed Group Mitoxantrone Hydrochloride 18 mg/m^2 | Relapsed/Refractory Group Mitoxantrone Hydrochloride 12 mg/m^2 | Relapsed/Refractory Group Mitoxantrone Hydrochloride 14 mg/m^2 | Relapsed/Refractory Group Mitoxantrone Hydrochloride 16 mg/m^2 | Relapsed/Refractory Group Mitoxantrone Hydrochloride 18 mg/m^2 | Phase 2 Newly Diagnosed Group 18 mg/m^2 | Phase 2 Relapsed/Refractory Group 16 mg/m^2
All-Cause Mortality (participants affected / at risk) | 0/9 | 2/9 | 2/9 | 1/6 | 6/10 | 4/6 | 4/6 | 2/4 | 40/106 | 21/34
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/6 | 0/10 | 0/6 | 0/6 | 0/4 | 0/106 | 0/34
Other Adverse Events (participants affected / at risk) | 8/9 | 8/9 | 9/9 | 6/6 | 10/10 | 6/6 | 6/6 | 4/4 | 100/106 | 31/34
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Newly Diagnosed Group Mitoxantrone Hydrochloride 12 mg/m^2 (N=9) | Newly Diagnosed Group Mitoxantrone Hydrochloride 14 mg/m^2 (N=9) | Newly Diagnosed Group Mitoxantrone Hydrochloride 16 mg/m^2 (N=9) | Newly Diagnosed Group Mitoxantrone Hydrochloride 18 mg/m^2 (N=6) | Relapsed/Refractory Group Mitoxantrone Hydrochloride 12 mg/m^2 (N=10) | Relapsed/Refractory Group Mitoxantrone Hydrochloride 14 mg/m^2 (N=6) | Relapsed/Refractory Group Mitoxantrone Hydrochloride 16 mg/m^2 (N=6) | Relapsed/Refractory Group Mitoxantrone Hydrochloride 18 mg/m^2 (N=4) | Phase 2 Newly Diagnosed Group 18 mg/m^2 (N=106) | Phase 2 Relapsed/Refractory Group 16 mg/m^2 (N=34)
Febrile Neutropenia (Infections and infestations) | 7 | 7 | 7 | 5 | 7 | 6 | 6 | 4 | 90 | 31
Fever (Infections and infestations) | 4 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 6 | 1
Tumor Lysis Syndrome (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 1 | 7 | 3
Maculopapular Rash (Skin and subcutaneous tissue disorders) | 2 | 2 | 6 | 1 | 2 | 2 | 0 | 1 | 27 | 3
Bacteremia (Infections and infestations) | 4 | 5 | 5 | 2 | 7 | 3 | 5 | 2 | 41 | 15
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 2 | 3 | 0 | 0 | 3 | 27 | 6
Fungal Pneumonia (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 22 | 5
Pneumonia (Infections and infestations) | 3 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 20 | 1
Cytokin Storm (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaphylaxis (Immune system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Papulopustular Rash (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 10 | 3
Soft Tissue Infection (Infections and infestations) | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 1 | 12 | 4
Catheter Related Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Skin Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 0 | 1 | 0 | 1 | 5 | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 8 | 0
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2 | 1 | 2 | 1 | 6 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 2
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Chloecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 2
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 11 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 6 | 3
Restrictive cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 6 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1
Intracranial hemorrhage (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0
Unequal limb length (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 7 | 2
Hepatic failure (Hepatobiliary disorders) | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 9 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 8 | 3
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 2
Vitreous hemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Multi-organ failure (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 3 | 0
Uveitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-04-17): https://cdn.clinicaltrials.gov/large-docs/96/NCT02044796/Prot_SAP_ICF_000.pdf